CLINICAL TRIAL: NCT05564234
Title: Role of Laparoscopy in Assessing Tumor Resectability in Ovarian Cancer Cases
Brief Title: Role of Laparoscopy in Assessing Resectability of Ovarian Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Muhannad Mohamed Elsayed Abdelrahman Azab, principle investigator, Zagazig University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: laparoscopy in ovarian cancer
Record Dates: First submitted 2022-09-26; First posted 2022-10-03 (Actual); Last update posted 2022-10-04 (Actual); Status verified 2022-10

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neoadjuvant chemotherapy (Active Comparator): cases with predictive index value score 8 or greater in which primary cytoreductive surgery was not feasible were were referred for neoadjuvant chemotherapy then interval cytoreductive surgery was done
  Interventions: Procedure: laparoscopy then neoadjuvant chemotherapy followed by interval cytoreductive surgery
- primary cytoreductive surgery (Active Comparator): cases with predictive index value score less than 8 were offered primary cytoreductive surgery.
  Interventions: Procedure: laparoscopy then primary cytoreductive surgery

INTERVENTIONS:
Procedure: laparoscopy then primary cytoreductive surgery — Laparoscopy was used to calcautation of fagotti PIV score , if less than 8 primary cytoreductive surgery were done.
  Arms: primary cytoreductive surgery
Procedure: laparoscopy then neoadjuvant chemotherapy followed by interval cytoreductive surgery — Laparoscopy was used to calcautation of fagotti PIV score and provides the histological diagnosis , if score more than 8 the patient were received neoadjuvant chemotherapy followed by interval cytoreductive surgery
  Arms: Neoadjuvant chemotherapy

SUMMARY:
Aim of Work is Prevention of unnecessary laparotomies and failed attempts to perform optimal cytoreduction in women with advanced ovarian cancer.

DETAILED DESCRIPTION:
Ovarian cancer is diagnosed at advanced stages in 80% of cases, leading to 5-year survival of approximately 30 %. Tumor reductive surgery and platinum and taxane-based chemotherapy has been the mainstay of treatment for advanced disease . The presence of residual disease after primary debulking surgery is a highly significant prognostic factor in women with advanced ovarian cancer. In up to 60 % of women, residual tumor of >1 cm is left behind after primary debulking surgery. These women might have benefited from neoadjuvant chemotherapy (NACT) prior to interval debulking surgery instead of primary debulking surgery followed by chemotherapy. Previous studies have demonstrated a clear survival benefit if resection to no gross residual disease (R0 resection) can be achieved, More extensive surgical procedures have been performed to achieve R0 status and have been associated with increased surgical morbidity. Accurate assessment of tumor burden at initial diagnosis using preoperative computed tomography, serum CA 125, and clinical factors has been used in models with variable success and has been difficult to standardize across surgical practices. It is important to determine at the time of diagnosis which patients should undergo primary tumor reductive surgery (TRS), and which should receive neoadjuvant chemotherapy (NACT) in order to minimize surgical morbidity and maximize the extent of cytoreduction. As such, several algorithms to predict the extent of disease encountered at cytoreductive surgery have been developed and evaluated . Fagotti et al. (2008) developed a laparoscopic scoring algorithm comprised of seven parameters: omental caking, peritoneal carcinomatosis, diaphragmatic carcinomatosis, mesenteric retraction, bowel infiltration, stomach infiltration, and liver metastases. . A laparoscopy-based scoring model developed by Fagotti et al.,(2008) demonstrated that a predictive index value score of 8 or greater had a specificity of 100%, positive predictive value of 100%, and negative predictive value of 70% for predicting a suboptimal primary tumor reductive surgery. Optimal tumor reductive surgery was defined as

1 cm or less in this model . Follow-up studies have demonstrated that laparoscopic scoring carries a low risk of complications; helps avoid unnecessary laparotomies in patients in whom cytoreduction to no gross residual disease would not be possible. To provide a more standardized approach to the management of patients with advanced ovarian cancer, this study will be performed to triage appropriate patients to laparoscopic scoring assessment using the previously validated scoring algorithm as reported by Fagotti, We will estimate the effects of the laparoscopic scoring algorithm in patients with advanced ovarian cancer to improve complete gross surgical resection rates and to determine the resulting clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with suspicious ovarian cancer by clinical and radiological assessment are included in this study.

Exclusion Criteria:

* Patients with poor Eastern Cooperative Oncology Group grade more than 2.
* Medical comorbidities at the time of diagnosis precluding primary surgery, newly diagnosed deep venous thrombosis or pulmonary embolus within 6 weeks of presentation.
* Immobile pelvic tumor reaching to xiphisternum leading to conclusions that complete cytoreductive surgery is not feasible
* Intrahepatic metastatic disease of more than one centimetre
* Para-aortic lymphadenopathy larger than one centimetre above the level of the renal veins
* Any contraindication for laparoscopy as cardiopulmonary compromise, intracranial diseases or large ventral hernia.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-12-09 (Actual); Primary Completion 2021-12-09 (Actual); Study Completion 2022-04-09 (Actual)

PRIMARY OUTCOMES:
complete gross resection of tumor | baseline
  The primary outcome for our study included improving complete gross resection rates at tumour cytoreductive surgery compared to historical data and avoids futile laparotomy defined as residual tumour with a maximum diameter more than 1 cm after primary cytoreductive surgery.

SECONDARY OUTCOMES:
Comparison between the accuracy of laparoscopy and CT with contrast on the abdomen | baseline
  The secondary outcomes included comparison between laparoscopic assessment and preoperative CT with contrast according to the accuracy of detection of
  * Omental lesion.
  * Peritoneal nodules.
  * Implantations on the surface of diaphragm.
  * Affection and retraction of the mesentry of bowel.
  * Intestinal infiltration.
  * Stomach implants.
  * Metastasis on hepatic or splenic surfaces.
surgical morbidity. | 1 month
  any complication during surgery or postoperative morbidity

CONTACTS AND LOCATIONS:
Overall Officials: wael hu elbrombly, MD, Study Director — faculty of medicine,zagazig univeristy; hanan at ghaly, MD, Study Director — faculty of medicine,zagazig univeristy; mohamed ab lashin, MD, Study Director — faculty of medicine,zagazig univeristy; muhannad mo azab, Msc, Principal Investigator — faculty of medicine,zagazig univeristy
Locations (1):
- Faculty of Medicine, Zagazig Univeristy, Zagazig, Sharqia Province, Egypt

REFERENCES:
- [Background] Fagotti A, Ferrandina G, Fanfani F, Ercoli A, Lorusso D, Rossi M, Scambia G. A laparoscopy-based score to predict surgical outcome in patients with advanced ovarian carcinoma: a pilot study. Ann Surg Oncol. 2006 Aug;13(8):1156-61. doi: 10.1245/ASO.2006.08.021. Epub 2006 Jun 21. PMID 16791447
- [Background] Fagotti A, Ferrandina G, Fanfani F, Garganese G, Vizzielli G, Carone V, Salerno MG, Scambia G. Prospective validation of a laparoscopic predictive model for optimal cytoreduction in advanced ovarian carcinoma. Am J Obstet Gynecol. 2008 Dec;199(6):642.e1-6. doi: 10.1016/j.ajog.2008.06.052. Epub 2008 Sep 17. PMID 18801470
- [Background] Fleming ND, Nick AM, Coleman RL, Westin SN, Ramirez PT, Soliman PT, Fellman B, Meyer LA, Schmeler KM, Lu KH, Sood AK. Laparoscopic Surgical Algorithm to Triage the Timing of Tumor Reductive Surgery in Advanced Ovarian Cancer. Obstet Gynecol. 2018 Sep;132(3):545-554. doi: 10.1097/AOG.0000000000002796. PMID 30095787